CLINICAL TRIAL: NCT06897826
Title: Acute Effect of Hamstring Stretching Performed With Proprioceptive Neuromuscular Facilitation Technique on the Endurance of Neck Deep Flexor Muscles in Healthy Women
Brief Title: Effect of Hamstring Stretching on Cervical Flexor Muscle Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ömer Osman Pala, associate professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AIBU-FTR-09
Record Dates: First submitted 2025-02-25; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Deep Neck Flexors; Hamstrings; Superficial Back Line; proprioceptive neuromuscular stimulation
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Group (Experimental): In this group participant's hamstring muscles stretched with PNF
  Interventions: Other: Proprioceptive neuromuscular facilitation
- Control Group (No Intervention): No application was made to this group

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation — The reason for choosing the proprioceptive neuromuscular facilitation technique is that it increases the hip flexion angle more than static stretching. Participants first lay down on the stretcher in a supine position. Then, the participant's lower extremity was lifted straight until the physiotherapist felt resistance. After reaching this position, the participant was asked to try to extend his lower extremity straight with half of his strength. After 10 seconds, the participant was given time to relax and after the participant relaxed, the lower extremity was brought to the new range of motion. This process was applied 3 times.
  Arms: PNF Group

SUMMARY:
The superficial posterior line is one of the eight main fascial lines defined on the body. One of the important muscle groups on this line is the hamstring muscle group. Studies have shown that various stretching methods applied to the hamstring muscle group affect the cervical region both in terms of range of motion and posture. As a result of this study, it was shown that deep neck flexor endurance increased in women who applied the PNF hold-relax method.

DETAILED DESCRIPTION:
The superficial posterior line is one of the eight main fascial lines defined on the body. One of the important muscle groups on this line is the hamstring muscle group. Studies have shown that various stretching methods applied to the hamstring muscle group affect the cervical region both in terms of range of motion and posture. Our aim in our study is to examine the effect of the proprioceptive neuromuscular stretching (PNF) method applied to the hamstring muscle group on the endura of the deep neck flexors based on these data.

ELIGIBILITY:
Inclusion Criteria:

* being female
* being healthy in musculoskeletal conditions

Exclusion Criteria:

* being hypermobile

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female people are eligible to participate for our study
Enrollment: 66 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Deep Neck Flexor Before and After | Two times in one day (before intervention, immediately after intervention)
  Deep neck flexor endurance changes before and after PNF hamstring stretch

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Osman PALA, phd, Study Director — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No